CLINICAL TRIAL: NCT01489397
Title: Magnified Intelligence Chromoendoscopy Plus Probe-based Confocal Laser Endomicroscopy for Gastric Intestinal Metaplasia Diagnosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Chulalongkorn Memorial Hospital (Other)
Responsible Party: Principal Investigator, Rapat Pittayanon, MD, Principle investigator, King Chulalongkorn Memorial Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RP002
Record Dates: First submitted 2011-12-05; First posted 2011-12-09 (Estimated); Last update posted 2014-06-11 (Estimated); Status verified 2014-06

CONDITIONS: Gastric Intestinal Metaplasia
Keywords: Confocol laser endomicroscopy; Feasibility of Confocol laser endomicroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gastric intestinal metaplasia (Experimental)
  Interventions: Device: Confocol laser endomicroscopy
- Normal (Placebo Comparator)
  Interventions: Device: Confocol laser endomicroscopy

INTERVENTIONS:
Device: Confocol laser endomicroscopy — Confocal laser endomicroscopy was applied at suspected lesion and normal mucosa followed by biopsy for pathology.

SUMMARY:
Magnified intelligence chromoendoscopy (FICE) plus probe-based confocal laser endomicroscopy (pCLE) for Gastric Intestinal Metaplasia (GIM) diagnosis: a feasibility trial

Research Question:

Is confocal endomicroscope feasible to diagnose gastric intestinal metaplasia?

Objective:

To evaluate the feasibility of confocal endomicroscope in diagnose gastric intestinal metaplasia.

Hypothesis:

Confocal endomicreosocpe can provide the accurate diagnosis of gastric intestinal metaplasia.

Research design:

Diagnostic study

Sample size:

The investigators follow the population in recent study from Imraporn et al.: Validity of magnify NBI for gastric intestinal metaplasia targeted biopsy (N= 50)

Data analysis:

Confocal Barrett's esophagus classification was used to evaluate agreement of confocal endomicroscopic finding in gastric intestinal metaplasia. The accuracy of new criteria for GIM by confocal endomicroscope was evaluated in relation to pathological report, a gold standard for diagnosis, and reported as sensitivity, specificity, positive predictive value, negative predictive value and accuracy of these criteria.

Expected Benefit and Application:

The feasibility of confocal endomicroscopy for diagnosis gastric intestinal metaplasia in order to improve the quality of GIM/dysplasia/early gastric cancer detection and then decrease the mortality rate from gastric cancer in the future.

DETAILED DESCRIPTION:
Background and Rationale:

Gastric cancer is the second leading cause of cancer related death in the world in recently data. The incidence and mortality rate is predominant in East Asia. Usually, gastric cancer is asymptomatic in early stage; therefore; most patients is in the advanced stage and incurable at diagnosis. The pathogenesis of intestinal type gastric cancer is sequential and multistep pathway. Moreover, the direction of pathway is irreversible beyond dysplasia. The equipment and/or procedure which can detect gastric dysplasia are very beneficial.

The recent study, Imraporn B et al., showed that narrow-banded imaging with magnification (NBI-ME) had a better sensitivity for gastric intestinal metaplasia (GIM) detection than a standard white light endoscopy (73% VS. 13%) and could detect two early gastric cancer from tissue pathology in 1-year follow-up cohort study. However, NBI-ME cannot differentiate among GIM, dysplasia and gastric cancer.

Confocal endomicroscope is a powerful instrument for performing high-resolution (x1,000 time) imaging to enable real-time histology and/or optical biopsy at the time of endoscopic examination(in vivo histology).Fluorescein, is a slightly acidic and hydrophilic dye, will be used as staining substance via IV administration. The fluorescein established a stable distribution throughout surface epithelial cells, which is regular columnar epithelium with round gland openings and cobblestone pattern; the connective tissue matrix of lamina propria; blood vessels, which are regular shape visible in the deeper mucosa; and red blood cells.It is not highly miscible with mucins, hence, mucins in goblet cells, which indicated GIM, will appear dark.

Because GIM is characterized by the diminutive lesions or microscopic abnormalities amidst large fields of diffuse disease, biopsy targeting and adequate sampling can be difficult and time consuming. Therefore, the instant resection with confocal microendoscope is not possible.

Consequently, the patient must be diagnosed GIM via a targeted NBI-ME biopsy first. And then endoscopic mucosal resection (EMR) via confocal endomicrosocpe is possible to be the complete therapeutic treatment for early gastric cancer within the same session at the suspected area of gastric dysplasia or neoplasia.

However, no study about confocal endomicroscope related early detection of gastric cancer was observed.

In this study, we must apply the endomicroscope's criteria from confocal Barrett's esophagus classification to indicate gastric dysplasia or neoplasia. The aim of this study is to evaluate the feasibility of confocal endomicroscopy to diagnose gastric intestinal metaplasia.

Review of related literature:

Confocal endomicroscope is available in 2005. The difference between white light endoscope and confocal endomicroscope.

Nowadays, a point-scanning fiber-optic fluorescein confocal endomicroscope for evaluate cellular morphology of the upper- and the lower-GI tract is possible. However, the improvement of diagnostic yield is evaluated in only Barrett's esophagus, colorectal cancer, detecting Helicobacter pylori. There is no exactly study about early detection of gastric cancer with confocal endomicroscope. Investigator use the confocal Barrett's esophagus classification to predict the area of dysplasia or neoplasia in stomach.

Assumption:

All patients have to undergo a targeted NBI-ME biopsy and never be treated as gastric cancer before.

Key Words:

Confocal endomicroscope Gastric intestinal metaplasia

Operational definition:

Gastric intestinal metaplasia/dysplasia/neoplasim is base on the updated Sydney classification.

Research methodology:

Population and Sample Target and sample population: The patients who were diagnosed gastric intestinal metaplasia (GIM) in the past 2 years in KCMH.

Observation and Measurement:

Collect the geographic data by interview and review the outpatient record. Evaluate the tissue pathology by one pathologist

Methodology:

1. All patients had informed the consent.
2. Take the history, physical examination and then fill in the record form
3. Set confocal endomicroscopy

   * 10% Fluorescein sodium 10 ml was injected intravenously.
   * 2.5-5 milligrams of intravenous midazolam and 10 milligrams of hyoscine were injected to sedate and decrease bowel movement for easier and complete visualization.
   * Simethicone solution was rinsed to reduce mucous and gas bubble in the stomach.
   * FICE was used to identify the area of suspected GIM.
   * Confocal endomicroscopy was performed and targeted to the suspected area. One snapshot images was recorded at the area of suspected and record the criteria of diagnosis GIM. Endoscopic resection was done at the suspected area.
   * DVD was recorded during the endoscopy.
4. Record the duration and complication of the procedure
5. Send the tissues to one clinically-blinded GI pathologist
6. Compare the pathology report and endoscopic finding
7. Report the result

Data collection:

All data are processed and recorded by one physician.

Ethical considerations:

There is not a clearly evidence about the serious side effect of fluorescein injection. If the patients had side effects during the research, the procedure will be terminated and the patients will be take care from KCMH staff.

Limitation:

This is a novel diagnostic tool to analyze living cells during endoscopy, especially for gastric intestinal metaplasia (GIM). There is not a standard criterion about confocal endomicroscopy finding in GIM. Investigator have to apply from Barrett's esophagus criteria and learn about criteria in GIM and gastric cancer.

Obstacles and strategies to solve the problems:

Because this is the study which base on the population from previous study by Imraporn et al., maybe some patients will loss follow up. The strategies to solve the problems are

1. Early call back to make an appointment
2. Collect new patients from the database of pathology department, KCMH

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 year-old
2. All patients were diagnosed GIM in the past 2 years.
3. All patients have to sign the consent form

Exclusion Criteria:

1. Previous gastric surgery including gastrectomy and bypass surgery
2. Bleeding tendency including decompensated cirrhosis, chronic kidney disease and long-tem antiplatelets or anticoagulants
3. Pregnanacy
4. History of fluorescein allergy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2010-04; Primary Completion 2011-12 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
The feasibility of confocal endomicroscope in diagnose gastric intestinal metaplasia | Up to 2 years
  If GIM can be detected properly, early gastric cancer(EGC) will be in early recognition. EGC can be cured by endoscopic resection and then the mortality rate from gastric cancer will be decrease.

CONTACTS AND LOCATIONS:
Locations (1):
- Rapat Pittayanon, Bangkok, Bangkok, Thailand

REFERENCES:
- [Derived] Pittayanon R, Rerknimitr R, Wisedopas N, Ridtitid W, Kongkam P, Treeprasertsuk S, Angsuwatcharakon P, Mahachai V, Kullavanijaya P. Flexible spectral imaging color enhancement plus probe-based confocal laser endomicroscopy for gastric intestinal metaplasia detection. J Gastroenterol Hepatol. 2013 Jun;28(6):1004-9. doi: 10.1111/jgh.12185. PMID 23432088
- See also: Related Info — http://www.medchulairb.com